CLINICAL TRIAL: NCT03476876
Title: Comparative Effectiveness of Two Acellular Matrices (Dermacell vs. Integra) for Management of Deep Diabetic Foot Ulcers - A Randomized Clinical Trial
Brief Title: Comparative Effectiveness of Two Acellular Matrices (Dermacell vs. Integra) for Management of Deep Diabetic Foot Ulcers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: LifeNet Health (Industry)
Responsible Party: Principal Investigator, Bijan Najafi, PhD, Professor of Surgery, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-42282
Record Dates: First submitted 2018-03-07; First posted 2018-03-26 (Actual); Results first posted 2023-07-07 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-06

CONDITIONS: Diabetic Foot Ulcer; Deep Diabetic Foot Ulcer
Keywords: acellular matrix
MeSH Terms: conditions — Diabetic Foot | interventions — integra artificial skin

STUDY DESIGN:
Intervention Model Description: The investigators will randomize using 1-1 ratio and based on diabetic foot ulcer cases. In the case that a subject had two eligible wound cases, the randomization will be done to have similar probably for the wound location (e.g. forefoot, mid-foot, hind-foot, etc). If an eligible subject had more than two wounds, only one of them will be considered as an intervention and only one of them as a control case.
Who Masked: Participant
Masking Description: Both of acellular dermal matrices are considered as a standard of care for non-healing diabetic foot ulcers. The subject will be unaware of type of matrices.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Dermacell (Experimental): Subject will receive treatment for one non-healing deep diabetic foot ulcer using one Dermacell acellular matrix. Subject will be followed up to 16 weeks post treatment, or until wound has closed, whichever comes first.
  Interventions: Combination Product: Dermacell
- Integra (Active Comparator): Subject will receive treatment for one non-healing deep diabetic foot ulcer using one Integra bilayer cross-linked matrix. Subject will be followed up to 16 weeks post treatment, or until wound has closed, whichever comes first.
  Interventions: Combination Product: Integra

INTERVENTIONS:
Combination Product: Dermacell — Subject will receive treatment for one non-healing deep diabetic foot ulcer using one Dermacell acellular matrix. Subject will be followed up to 16 weeks post treatment, or until wound has closed, whichever comes first.
  Other Names: Dermacell acellular dermal matrix placed in one lesion
  Arms: Dermacell
Combination Product: Integra — Subject will receive treatment for one non-healing deep diabetic foot ulcer using one Integra bilayer cross-linked matrix. Subject will be followed up to 16 weeks post treatment, or until wound has closed, whichever comes first.
  Other Names: Integra bilayer cross-linked matrix placed in one lesion
  Arms: Integra

SUMMARY:
Diabetes-related foot ulcers (DFUs) are a leading cause of hospitalization and amputation worldwide, and account for 33% of all direct costs of diabetes care in the US. Ulcers requiring acute care can result in treatment costs of up to US$70,000 per event, varying with the severity of the wound. Once the skin is ulcerated, it is susceptible to becoming infected and ultimately amputation in particular in case of deep DFUs. To manage the cost and avoid hospitalization and amputation, wound should be immediately closed. But this is often challenging in diabetic foot with deep ulcers.Wound healing is a dynamic process involving interactions between cells, extracellular matrix (ECM) and growth factors that reconstitutes tissue following injury. ECM plays an important role in tissue regeneration and is the major component of the dermal skin layer. Recognition of the importance of the ECM in wound healing has led to the development of wound products that aim to stimulate or replace the ECM in particular in case of deep tissue destruction because of deep DFUs. It is known from the literature that chronic or hard-to-heal wounds are characterized by a disrupted or damaged ECM that cannot support wound healing. Thus treatment strategies based on use of biologic scaffold materials for management of chronic and deep wounds has increased dramatically during the past two decades. These scaffolds include those comprising an intact extracellular matrix (ECM) or individual components of the ECM, and those comprising hybrids incorporating a synthetic component with a biologic component. DermACELL (LifeNet Health,Virginia Beach, VA) is acellular dermal matrices (ADM), which has been shown to be effective in treating chronic DFUs in a clinical trial.

Another ADM product available in the market is made by Integra® (Bilayer Matrix Wound Dressing, Integra LifeSciences). However, advantages/disadvantages of one compared to the other are unclear. In addition, prior studies often focused on wound healing outcomes (e.g. time to heal, success of wound healing) without considering patient-centered and physician-centered outcomes such as time and difficulty to apply, likelihood of adverse events and need for reapplication, poor tissue mechanics outcomes (e.g. presence of scarring or tissue biomechanics properties leading to increase in shear or pressure post healing thus increasing likelihood of recurrence of the ulcer), and other patient centered outcomes like smell, pain, and comfort.

The primary objective of this prospective, randomized trial is to compare the outcomes of DermaCELL with Integra. The investigators assumed that the wounds outcomes (e.g. weekly wound size change, time to heal, time to successful wound granulation) are comparable between DermaCELL and Integra. However, from operation and patient centered outcomes, there may be some noticeable differences. For instance, DermaCELL, thanks to its mesh structure, thin thickness, and no need for hydration, may be easier to apply with shorter time than Integra. The factors are of key importance in operation room (OR) setting and could reduce overall cost of application and needs in using OR resources. Other important outcomes least addressed in prior studies are number of grafts failing, adverse events (e.g. amputation, infection, etc), cost of wound healing treatment, tissue biomechanics, which may lead to recurrence of ulcers (e.g. formation of tissue scarring), and other patient-centered outcomes (e.g. pain, quality of sleeping, wound smelling, etc). For instance, many patients are unhappy with smelling of wounds, which make them embarrassed among their family members like grand kids. Thus reducing wound smelling during activities of daily living is often considered as an important patient centered outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Non-infected deep wounds (Grade 2 Wagner Ulcer Classification)

Exclusion Criteria:

* Minors
* Wounds with bone exposure
* Active infection
* Gangrene or osteomyelitis
* Major vascular problems (ABI <0.5 or >1.3)
* Unable to comply with follow up visits (e.g. long distance travel)
* Unable or unwilling to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2021-04-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: lesions
Groups:
- Dermacell: Subject will receive treatment for one non-healing deep diabetic foot ulcer using one Dermacell acellular matrix. Subject will be followed up to 16 weeks post treatment, or until wound closure, whichever comes first.
- Integra: Subject will receive treatment for one non-healing deep diabetic foot ulcer using Integra bilayer cross-linked matrix. Subject will be followed up to 16 weeks post treatment, or until wound closure, whichever comes first.
Period: Overall Study
Arm/Group | Dermacell | Integra
Started | 19; 19 lesions | 15; 15 lesions
Completed | 9; 9 lesions | 7; 7 lesions
Not Completed | 10; 10 lesions | 8; 8 lesions

BASELINE CHARACTERISTICS:
Population: All baseline data were collected on the participant level
Groups:
- Participants Receiving Dermacell Acellular Dermal Matrix in One Lesion: Subject will receive treatment for one non-healing deep diabetic foot ulcer using one Dermacell acellular dermal matrix. Subject will be followed up to 16 weeks post treatment, or until the wound has closed, whichever comes first.
- Participants Receiving Integra Bilayer Cross-linked Matrix in One Lesion: Subject will receive treatment for one non-healing deep diabetic foot ulcer using one Integra bilayer cross-linked matrix. Subject will be followed up to 16 weeks post treatment, or until wound has closed, whichever comes first.
- Total: Total of all reporting groups
Arm/Group | Participants Receiving Dermacell Acellular Dermal Matrix in One Lesion | Participants Receiving Integra Bilayer Cross-linked Matrix in One Lesion | Total
Number analyzed (Participants) | 19 | 15 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 11 | 25
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.5 (10.1) | 56.6 (13.5) | 59 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 7 | 12 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 5 | 11
  White | 11 | 9 | 20
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Wound Area at 16 Weeks
Description: Wound area in squared centimeters will be quantified using Aranz Medical Image processing system. The wound will be manually traced using Aranz Medical to obtain length and width. Then the average of wound per group will be compared at 16 weeks.
Time Frame: An average of 16 weeks.
Population: one lesion per subject was analyzed. Data from 18 subjects was unable to be collected at last follow up visit due to drop out of the study.
Measure: Mean (Standard Deviation); unit: cm^2
Units Other Than Participants: lesions
Arm/Group | Dermacell | Integra
Number analyzed (Participants) | 9 | 7
Number analyzed (lesions) | 9 | 7
cm^2 | 6.1 (6.5) | 6.8 (8)

2. Primary Outcome: Percentage of Wound Granulation at 16 Weeks
Description: Percentage of wound granulation will be subjectively assessed based on the observation and criteria of the treating clinician. After cleaning the wound, the clinician will provide with a percentage of granulated tissue based on his/her observation. Then, the average of wound granulation per group will be compared at 16 weeks
Time Frame: An average of 16 weeks.
Population: One lesion per participant will be analyzed. Data from 18 subjects was unable to be collected due to drop out of the study.
Measure: Mean (Standard Deviation); unit: percentage of wound granulation
Units Other Than Participants: lesions
Groups:
- Integra: Subject will receive treatment for one non-healing deep diabetic foot ulcer using one Integra bilayer cross-linked matrix. Subject will be followed up to 16 weeks post treatment, or until wound closure, whichever comes first.
Arm/Group | Dermacell | Integra
Number analyzed (Participants) | 9 | 7
Number analyzed (lesions) | 9 | 7
percentage of wound granulation | 80.44 (31.5) | 96.7 (5.1)

3. Primary Outcome: Lower Extremity Skin Perfusion at 16 Weeks
Description: Skin perfusion will be quantified by Skin Perfusion Pressure Test (SPP) using Sensilase PAD-IQ (VASAMED) on the lower extremities. This tests utilizes a cuff with sensors placed above the ankle level which measures the lower extremity distal skin perfusion pressure in millimeters of mercury (mmHg) while eliciting and releasing pressure to the vasculature of the lower leg through the cuff. Then, the average of mmHg per group will be compared at 16 weeks.
Time Frame: An average of 16 weeks.
Population: One leg (which contains the lesion) per patient was analyzed. Data from 18 subjects was unable to be collected due to drop out of the study. Data from the resting 14 subjects was unable to be collected at last follow up visit due to patient comfortability, lower extremity manipulation, risk for infection, or device component (sensors) discontinuation.
Measure: Mean (Standard Deviation); unit: mmHg
Units Other Than Participants: legs
Arm/Group | Dermacell | Integra
Number analyzed (Participants) | 2 | 0
Number analyzed (legs) | 2 | 0
mmHg | 62.5 (13.4) |

4. Primary Outcome: Wound Saturation of Oxygen at 16 Weeks
Description: Wound saturation of oxygen will be quantified using Near Infrared Spectroscopy by Kent Imaging system. Kent is a non-invasive camera that detects wound saturation of oxygen with a simple spectral picture. After taking the picture, each wound will be traced allowing for accurate and detailed data collection. Then, the average of saturation of oxygen of wounds per group will be compared at 16 weeks.
Time Frame: An average of 16 weeks.
Population: One lesion per participant was analyzed. Data from 18 subjects was unable to collect due to drop out of study. Data from the resting 1 subject was unable to be collected at last follow up visit due to patient non-compliance.
Measure: Mean (Standard Deviation); unit: percentage of saturation of oxygen
Units Other Than Participants: lesions
Arm/Group | Dermacell | Integra
Number analyzed (Participants) | 8 | 7
Number analyzed (lesions) | 8 | 7
percentage of saturation of oxygen | 65.5 (22.8) | 83.1 (8.1)

5. Secondary Outcome: Number of Participants With Frailty
Description: Frailty assessment will be measured with the Trauma Specific Frailty Index (TSFI) score. The total score of 15 variables including cardiovascular and cognitive comorbidities, and features such as mobility assistance, mood status, physical function, and nutritional status will be taken into consideration to determine whether a patient is frail. The minimum score is 0 and the maximum score is 0.3. A total score (including the 15 variables) of >0.27 is considered as frail. A score of ≤0.27 score is considered as non-frail.
Time Frame: Only baseline, time of recruitment
Measure: Count of Participants; unit: Participants
Arm/Group | Dermacell | Integra
Number analyzed (Participants) | 19 | 15
Participants | 11 | 8

6. Secondary Outcome: Time of Graft Application to One Wound During Baseline Procedure
Description: Duration of graft application will be measured from the time of the graft being placed on the wound, to the time of the last suture/staple to secure the graft placement. Time will be counted in seconds. Then, the average of time per group will be compared to the other group.
Time Frame: Only at baseline, time of recruitment
Population: All patients received a graft at the study enrollment. Therefore, the average time of graft placement was obtained from all the subjects at baseline.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: grafts
Arm/Group | Dermacell | Integra
Number analyzed (Participants) | 19 | 15
Number analyzed (grafts) | 19 | 15
seconds | 879.1 (501.8) | 667.5 (561.4)

7. Secondary Outcome: Number of Participants With Graft Re-application to One Wound at 16 Weeks
Description: Number of participants in need to re-apply at least one same or different graft(s) to one wound in approximately 16 weeks
Time Frame: An average of 16 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Dermacell | Integra
Number analyzed (Participants) | 9 | 7
Participants | 3 | 0

8. Secondary Outcome: Number of Participants With Wound Complications at 16 Weeks
Description: Complication is described as infection, necrosis, bleeding, or graft-rejection of one wound per patient.
Time Frame: An average of 16 weeks.
Measure: Count of Participants; unit: Participants
Groups:
- Dermacell: Subject will receive treatment for non-healing deep diabetic foot ulcer using Dermacell acellular matrix. Subject will be followed up to 16 weeks post treatment, or until wound closure, whichever comes first.
- Integra: Subject will receive treatment for non-healing deep diabetic foot ulcer using Integra bilayer cross-linked matrix. Subject will be followed up to 16 weeks post treatment, or until wound closure, whichever comes first.
Arm/Group | Dermacell | Integra
Number analyzed (Participants) | 19 | 15
Participants | 10 | 8

ADVERSE EVENTS:
Time Frame: 16 weeks
Groups:
- Dermacell: Subject will receive treatment for deep diabetic foot ulcer using Dermacell acellular matrix. Subject will be followed up to 16 weeks post treatment, or until wound closure, whichever comes first.
  Dermacell: Subject will receive treatment for deep diabetic foot ulcer using Dermacell acellular matrix. Subject will be followed up to 16 weeks post treatment, or until wound closure, whichever comes first.
- Integra: Subject will receive treatment for deep diabetic foot ulcer using Integra acellular matrix. Subject will be followed up to 16 weeks post treatment, or until wound closure, whichever comes first.
  Integra: Subject will receive treatment for deep diabetic foot ulcer using Integra acellular matrix. Subject will be followed up to 16 weeks post treatment, or until wound closure, whichever comes first.
Arm/Group | Dermacell | Integra
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/15
Other Adverse Events (participants affected / at risk) | 0/19 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03476876/Prot_SAP_004.pdf
  • Informed Consent Form (2019-12-03): https://cdn.clinicaltrials.gov/large-docs/76/NCT03476876/ICF_005.pdf